CLINICAL TRIAL: NCT06353204
Title: The Evaluation of the Effectiveness of the Diversion Measure Halt-intervention: a Randomized Controlled Trial
Brief Title: Effectiveness of the Justice Diversion Halt-intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wetenschappelijk Onderzoek en Datacentrum (Other Government)
Collaborators: Utrecht University (Other); Leiden University (Other)
Responsible Party: Principal Investigator, André van der Laan, Prof. dr., Wetenschappelijk Onderzoek en Datacentrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3325
Record Dates: First submitted 2024-03-12; First posted 2024-04-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-04

CONDITIONS: Criminal Recidivism; Delinquency; Antisocial Behavior
MeSH Terms: conditions — Recidivism; Antisocial Personality Disorder

STUDY DESIGN:
Intervention Model Description: A comparison between two groups will be made. One half of the participants will be randomly assigned to a group that receives the Halt-intervention, while the other group receives no Halt-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Halt-intervention (Experimental): The experimental group will receive the Halt-intervention.
  Interventions: Behavioral: Halt-intervention
- Control group: No Halt-intervention (No Intervention): The control group will not receive the Halt-intervention, nor will they receive any other intervention or form of punishment.

INTERVENTIONS:
Behavioral: Halt-intervention — The Halt-intervention is a Dutch extrajudicial, or diversion, measure for minors (aged 12-17) who committed a minor offence. The intervention can consist of conversations with the Halt-employee, working or learning assignments to learn from the mistakes made or to work on certain skills, such as social skills, and/or apologizing to the victim.
  Arms: Experimental group: Halt-intervention

SUMMARY:
In the current study the effectiveness of the Dutch diversion measure Halt is investigated using a randomized controlled trial. Because of the thorough scientific substantiation of the intervention theory, it is hypothesized that receiving the Halt-intervention will lead to less recidivism in comparison to receiving no intervention.

DETAILED DESCRIPTION:
The Halt-intervention is a widely used Dutch diversion measure for youth (aged 12-17) who committed a minor offence. In the current study, it will be investigated whether the Halt-intervention is successful in reducing recidivism and in achieving the intervention goals. The effectiveness will be assessed using a randomized controlled trial. Participants will be randomly assigned to the experimental condition in which participants will receive the halt intervention or to the control condition in which participants will not receive an intervention. Participants fill out three self-reported questionnaires over a time period of one year. With these questionnaires is it investigated whether the intervention is successful in achieving the different intervention goals (improving social skills, taking responsibility, correct wrongdoing or damage, improving conventional beliefs and improving support from the social network) and in achieving a reduction in recidivism. Furthermore, the adherence to children's rights in the practice of Halt is investigated. Lastly, two years after the first contact with Halt recidivism is assessed using official police and judicial records.

ELIGIBILITY:
Inclusion Criteria:

* Juveniles who have been referred to Halt after committing a minor offence that is eligible for the Halt-intervention.
* Juveniles between the ages of 12 and 18.

Exclusion Criteria:

* Participants who do not speak Dutch or who do not speak Dutch fluently.
* Participants who have already participated in the study before.
* Participants who are participating in the following Halt-programs: 'Hack_right', 'Respect Online' or 'Sport en Spel'.
* Participants of whom it is suspected that their are serious concerns for their safety.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Criminal Recidivism based on self-report | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  Assessed using the items from the Youth Delinquency Survey.
Criminal Recidivism based on official police records | T3 (24 month follow up)
  Assessed using official Dutch Police registration records.
Criminal Recidivism based on official judiciary records | T3 (24 month follow up)
  Assessed using official Dutch judicial records.
Truancy based on self-report | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  Assessed using the items from the Youth Delinquency Survey.

SECONDARY OUTCOMES:
Conventional beliefs | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  Self-reported degree of conventional beliefs, or attitude towards delinquency, assessed using the Dutch translation of the Attitudes Towards Delinquent Behavior (ATDS) questionnaire (translated by the WODC).
Minimizing/mislabeling | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree in which the consequences of delinquent behavior are minimized, mislabeled or seen as acceptable, assessed using the How I Think (HIT) subscale 'Minimizing/Mislabeling' using the Dutch translation ('Hoe Ik Denk (HID)).
Social skills | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree in which pressure from friends to conduct delinquent behavior is experienced, assessed using a (self-developed) Dutch translation of the Peer Pressure Scale.
Taking responsibility for the consequences of behavior | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree to which a sense of guilt, or responsibility, for the consequences for delinquent behaviour is experienced, assessed using the How I Think (HIT) subscale 'Blaming Others' using the Dutch translation ('Hoe Ik Denk' (HID)).
Correct wrongdoing | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree in which the wrongdoing and/or damages are corrected, assessed using a self-developed scale consisting of four question about having a conversation with the victim, apologizing to the victim, paying for the victim's damages and correcting the damages made.
Support from social network | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree in which support from the social network is experienced and the degree in which respondents experience that they can ask their social network for help or advise (for example friends and family). Assessed using the Multidimensional Scale of Perceived Social Support. Scale is translated to Dutch by the WODC.
Experienced legitimacy | T0 (baseline); T1 (100 days follow up)
  Experienced legitimacy during the first contact with Halt (experimental and control group) and during the Halt-intervention (experimental group), assessed using a four-item scale.
Experienced treatment | T0 (baseline); T1 (100 days follow up)
  Experienced treatment during the first contact with Halt (experimental and control group) and during the Halt-intervention (experimental group) by the Halt-employee, assessed using a seven-item scale.
Receiving adequate information | T0 (baseline); T1 (100 days follow up)
  The degree to which the information given during the first contact with Halt (experimental and control group) and during the Halt-intervention (experimental group) about the Halt-intervention is experienced as adequate and comprehensible, assessed using a self-developed six-item scale.
The right to be informed | T0 (baseline); T1 (100 days follow up)
  The degree to which participants have the feeling that they are heard during the first contact with Halt (experimental and control group) and during the Halt-intervention (experimental group), assessed using a self-developed six-item scale.
Experienced voluntariness | T0 (baseline); T1 (100 days follow up)
  The degree to which participants experience being forced to confess the crime they committed, assessed using a self-developed three-item scale. Participants are asked (1) whether they feel that they were forced to confess their crime, (2) whether they feel it is justified that they are referred to Halt and (3) whether they feel that it is their own choice to go to Halt. These items will be presented to participants in the experimental and control group during T0 and to participants in the experimental group during T1.
Access to legal assistance | T0 (baseline); T1 (100 days follow up)
  The degree to which participants have access to an attorney, assessed using two self-developed questions. Participants are asked whether they had the opportunity to (1) speak to a lawyer about their offence and had the opportunity to (2) speak to a lawyer about their referral to Halt. These items will be presented to participants in the experimental and control group during T0 and to participants in the experimental group during T1.
Knowledge of not obtaining a criminal record | T0 (baseline); T1 (100 days follow up)
  Whether or not participants are aware of the fact that completion of the Halt-intervention results in not obtaining a criminal record (yes/no). These items will be presented to participants in the experimental and control group during T0 and to participants in the experimental group during T1.
Experienced stigmatisation | T1 (100 days follow up); T2 (12 month follow up)
  The degree of experienced stigmatization, assessed using the four-item Stigmatisation subscale of the Re-integrative Shaming questionnaire.
Experienced re-integration | T1 (100 days follow up); T2 (12 month follow up)
  The degree of experienced re-integration, assessed using the four-item Re-integration subscale of the Re-integrative Shaming questionnaire.

OTHER OUTCOMES:
Mental health problems during the last six months | T0 (baseline)
  The degree to which risk and/or protective factors are present, assessed using the Strength and Difficulties Questionnaire (SGQ) using the Dutch translation.
Experienced problems | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  Experienced problems in different domains (at home, school, alcohol, money, drugs, health, mental health, gaming) and whether their has been professional help for these problems using the ten-item scale from the Youth Delinquency Survey.
Delinquent friends | T0 (baseline; T1 (100 days follow up); T2 (12 month follow up)
  The degree in which participants have delinquent friends, assessed using a six-item scale from the Youth Delinquency Survey.
Parental involvement | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The degree of parental control, parental monitoring and parental solicitation, assessed using the Dutch translation of the Parental Monitoring Questionnaire.
Demographical characteristics | T0 (baseline); T1 (100 days follow up); T2 (12 month follow up)
  The different demographical characteristics of respondents, such as gender and age.
Halt-intervention program integrity | T1 (100 days follow up)
  Questionnaire is being developed.
Characteristics Halt-employee | T1 (100 days follow up)
  Questionnaire is being developed.
Perceived relationship with Halt-employee | T1 (100 days follow up)
  Questionnaire is being developed.
Educational attainment | T1 (100 days follow up)
  The most recent completed type of education assessed using the registration system of the Halt-intervention. .
Type of criminal offense | T1 (100 days follow up)
  The type of criminal offense (e.g. shoplifting, petty theft) as registered in the registration system of the Halt-intervention.
Characteristics of referral to Halt-intervention | T1 (100 days follow up)
  The organisation that referred to Halt (police or truancy officer) assessed using the registration system of the Halt-intervention.
Types of modules used during the Halt-intervention | T1 (100 days follow up)
  The Halt-intervention contains of different modules, such as 'Handling Anger'; 'Handling Peer Pressure'; 'Making an apology to the victim'. These modules will be assessed using the registration system of the Halt-intervention.
Parts of the Halt-intervention carries out as group or solo intervention | T1 (100 days follow up)
  The Halt-intervention can be offered as a solo of as a group intervention. The different forms used are assessed using the registration system of the Halt-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: André M. van der Laan, Prod. Dr., Principal Investigator — Wetenschappelijk Onderzoek en Datacentrum
Locations (1):
- WODC, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study is part of a dissertation consisting of multiple articles which will be offered for publication to peer reviewed journals. First the study protocol article will be written and offered for publication to a peer reviewed journal, including a brief Statistical Analysis Plan (SAP) and as supplement the Informed Consent Form (ICF). Thereafter the study results articles will be offered for publication to peer reviewed journals asap. During this period there is no plan to make individual participant data (IPD) available.